CLINICAL TRIAL: NCT06187779
Title: Influence of Lower Segment Thickness on Induction of Labor With Balloon Insertion (ATAD)
Brief Title: Induction ATAD Catheter and Lower Segment Thickness
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MEIRATAD
Record Dates: First submitted 2023-12-17; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Induction of Labor Affected Fetus / Newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Segmental thickness measurement (Experimental): This population's lower segment will be measured.
  Interventions: Other: Lower segment measurment
- Segmental thickness no measurement (No Intervention): No measurements of lower segment.

INTERVENTIONS:
Other: Lower segment measurment — Lower segment measurement will be taken prior to induction with a balloon catheter (ATAD).
  Arms: Segmental thickness measurement

SUMMARY:
A prospective cohort study of pregnant women undergoing induction of labor at term .inculding- Women with a singleton pregnancy at ≥ 37 weeks' gestation, with a live fetus in cephalic presentation. all women will undergo transvaginal ultrasound assessment before induction of labor admission. Maternal and obstetric characteristics and Bishop score will be recorded. The main outcome is the overall rate of Cesarean delivery after induction of labor.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age above 24 weeks
* Singleton
* Vertex position
* Labor induction based on obstetrics guidelines

Exclusion Criteria:

* C/I for Induction of labor
* C/I for vaginal birth
* Multiple gestation
* Known fetal anatomical or genetic anomalies.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — For pregnant patient
Enrollment: 500 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2025-12-06 (Estimated); Study Completion 2026-12-06 (Estimated)

PRIMARY OUTCOMES:
Cesarean section prevalence | during labor
  Number of patients who delivered with CS

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel